CLINICAL TRIAL: NCT03559660
Title: Compassionate Use Program Certolizumab Pegol (CDP-870) in Adults Suffering From Crohn's Disease (CD)
Brief Title: CUP Certolizumab Pegol (CDP-870) in Adults Suffering From Crohn's Disease (CD)
Acronym: COMPAS
Status: No longer available | Type: Expanded Access
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: C87092
Record Dates: First submitted 2018-06-05; First posted 2018-06-18 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Certolizumab Pegol
  Other Names: Cimzia

SUMMARY:
The objective of this program is to allow treating physicians to supply/continue to supply Certolizumab Pegol (CIMZIA®, CZP) to adults suffering from Crohn's Disease (CD), and who are considered not suitable for treatment, intolerant, have medical contraindications or had insufficient response with an authorized conventional therapy, including other authorized biologics.

ELIGIBILITY:
Inclusion Criteria:

- Patient comes from ending open label studies such as WELCOME -C87046, COSPAR - C87065, MUSIC - C87043, PRECISE 3 - C87033, PRECISE 4 - C87034 and C87088

Exclusion Criteria:

* Patient has been treated with any experimental biological or non biological therapy other than Certolizumab Pegol (CZP) within 5 plasma half-lifes*
* Has been treated with an approved biological, namely infliximab within the last 8 weeks, and adalimumab within the last 2 weeks*
* Known hypersensitivity to CZP or any of its excipients
* Current or recent history of severe, progressive, uncontrolled renal, hepatic, haematological, gastrointestinal (other than Crohn's disease), endocrine, pulmonary, cardiac, neurological, or cerebral disease
* Serious or life threatening infection within the last 6 months, any signs of current or recent infection
* Active or latent tuberculosis (TB): if one or more of the 3 criteria is positive for evidence of TB infection*:

  1. A medical history of or a recent (< 6 months) active tuberculosis (TB)
  2. A recent (<6 months) chest X-ray with signs consistent with TB infection
  3. A recent (<6 months) positive purified protein derivative (PPD) skin test (defined as induration or 5mm or more) and/or an indeterminate or positive QuantiFERON-TB Gold or Elispot test.

It is recommended that patients are monitored at least annually for active and latent TB by both 1) a chest X-ray read by a pulmonologist or radiologist and 2) a PPD skin test and/or Elispot/ QuantiFERON TB Gold test

* Patient received live vaccinations including, but not limited to, oral polio, herpes zoster, measles-mumps-rubella (MMR) or nasal influenza within the last 8 weeks or has planned live immunizations during the planned period of administration of CZP
* Known prior or concurrent viral hepatitis B and C
* Known Human Immunodeficiency Virus (HIV) infection
* Concurrent malignancy or a history of malignant disease
* History of a lymphoproliferative disorder or any signs or symptoms suggestive of this disease
* History of, or suspected or confirmed active demyelinating disease of the central nervous system
* History of or concurrent New York Heart Association (NYHA) Class III/IV heart failure
* As the safety and efficacy of CZP has not been established in patients younger than 18 years of age, drug is not recommended for use in these patients until further data are available
* As no data are available in pregnant women, drug should not be administered to female patients of childbearing potential - unless an adequate method of contraception is used - or to pregnant/lactating female patients.*

'*' Not applicable (NA) for patients on treatment with CZP from trials such as WELCOME -C87046, COSPAR -C87065, MUSIC - C87043, PRECISE 3 - C87033, PRECISE 4 - C87034 and C87088.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)